CLINICAL TRIAL: NCT07044804
Title: Brain-directed Treatment to Improve Language in Adolescents and Young Adults With Down Syndrome: the Efficacy of Transcranial Direct Current Stimulation Coupled With Linguistic Training.
Brief Title: Non-Invasive Brain Stimulation to Improve Language in Down Syndrome.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Floriana Costanzo (Other)
Collaborators: Bambino Gesù Children's Hospital IRCCS (Other)
Responsible Party: Sponsor-Investigator, Floriana Costanzo, Psychologist, PhD, Bambino Gesù Hospital and Research Institute
Organization: Bambino Gesù Hospital and Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3406_OPBG_2024; Jérôme Lejeune Foundation (Other Grant/Funding Number: Jérôme Lejeune Foundation)
Record Dates: First submitted 2025-06-20; First posted 2025-07-01 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2024-08

CONDITIONS: Down Syndrome
Keywords: Trisomy 21; tDCS; Non-invasive brain stimulation; Speech; Neuroplasticity; BDNF; neurofilament light chain
MeSH Terms: conditions — Down Syndrome; Speech; Charcot-Marie-Tooth disease, Type 1F

STUDY DESIGN:
Intervention Model Description: This is a no profit, single center, prospective, randomized double-blind placebo controlled study to assess the superiority of tDCS active treatment to placebo. Enrollment will last 15 months, with the study expected to start in August 2024.Participants and evaluators will be blinded to treatment. Every tDCS session will be conducted during a language training in the Italian language, in order to optimize the intervention. A neuropsychological, linguistic, behavioural and functional communication assessment will be carried prior to (T0), following the end of the treatments (T1) and after three months (T2). Additional biological and neurophysiological measures will be collected. Specifically, the assessment of BDNF and NfL levels and EEG will be performed before and at the end of treatment, and at a 3 month after the end of treatment, to evaluate the involvement and changes in neuronal plasticity mechanisms in response to neuromodulation treatment and language training.
Who Masked: Participant, Outcomes Assessor
Masking Description: Both participants and evaluators will be blinded to the treatment conditions. To control for a possible placebo effect, the study included the control group placebo tDCS plus language training.
  It is well known that tDCS has a sham mode that cannot be easily detected by participants, making it possible to be used in controlled experiments and randomized controlled clinical trials. The opening of the blind will be allowed if serious adverse events occur or if the subject wants to leave the study early.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active Anodal tDCS to the left IFG (Active Comparator): Anodal- tDCS will be delivered by a battery driven, constant current stimulator through a pair of saline-soaked sponge electrodes kept firm by elastic bands. The device employed will be the BrainStim+ (REF: EMS BSTIM+), a lightweight, battery-operated constant current stimulator.The active electrode will be placed on the left IFG cortex (between F5 and F7 of the extended International 10-20 system for EEG electrode placement) cortex and the reference electrode placed above the contralateral shoulder, as previously applied in DS.Stimulation intensity will be set at 1 mA; the duration of stimulation will be 20 min and will be held five consecutive daily session per week for two weeks for a total of 10 sessions. During the tDCS sessions participant will sit in a comfortable chair and a language training will be administered for 20 minutes.
  Interventions: Device: Active Group (Active Anodal tDCS to the left IFG or Cathodal tDCS to the left IFG)
- Active Cathodal tDCS to the left IFG (Active Comparator): Cathodal- tDCS the cathode will be placed on the left IFG (between F5 and F7 of the extended International 10-20 system for EEG electrode placement) cortex, while the anode will be placed above the right shoulder. The device employed will be the BrainStim+ (REF: EMS BSTIM+), a lightweight, battery-operated constant current stimulator. Stimulation intensity will be set at 1 mA; the duration of stimulation will be 20 min and will be held five consecutive daily session per week for two weeks for a total of 10 sessions. During the tDCS sessions participant will sit in a comfortable chair and a language training will be administered for 20 minutes.
  Interventions: Device: Active Group (Active Anodal tDCS to the left IFG or Cathodal tDCS to the left IFG)
- Sham tDCS to the left IFG (Sham Comparator): In the sham condition, participants will undergone electrode placements identical to those used in either the anodal or cathodal tDCS configurations, with equal allocation to each montage. The BrainStim+ device (REF: EMS BSTIM+), a lightweight, battery-operated constant current stimulator, will be used. However, the current will be applied only briefly for 30 seconds before being ramped down in a manner imperceptible to the participant, thereby simulating the initial sensation of stimulation without delivering an active dose.
  Sham sessions will follow the same schedule as the active conditions-20 minutes per session, five consecutive daily sessions per week over two weeks (total of 10 sessions). During each session, participants will be seated comfortably and engage in concurrent language training.
  Interventions: Device: Sham Group

INTERVENTIONS:
Device: Active Group (Active Anodal tDCS to the left IFG or Cathodal tDCS to the left IFG) — Participants in the active tDCS group (Anodal tDCS or Cathodal tDCS) will receive stimulation set at 1 mA (milliampere), with a duration of 20 minutes per session. The stimulation will be administered in five consecutive sessions per day, five days a week, for two weeks, totaling 10 sessions, while participants will also undergo logopedic treatment for 20 minutes. The training protocol will consist of 10 minutes of training in motor planning and programming abilities and 10 minutes of training on the lexical, morphosyntactic, and functional aspects of language and communication.
  Arms: Active Anodal tDCS to the left IFG; Active Cathodal tDCS to the left IFG
Device: Sham Group — For the sham condition, the same electrode placement will be used as in the anodal tDCS condition, but the current will be applied for 30 s and will be ramped down without the participant's awareness. Stimulation intensity will be set at 1 mA; the duration of stimulation will be 20 min and will be held five consecutive daily session per week for two weeks, for a total of 10 sessions. During the tDCS sessions participant will sit in a comfortable chair and a language training will be administered
  Arms: Sham tDCS to the left IFG

SUMMARY:
Down syndrome (DS) is associated with cognitive deficits, caused by alterations in neuroplasticity and synaptic transmission. Non-invasive brain stimulation techniques, such as transcranial direct current stimulation (tDCS), can modulate the brain's plasticity mechanisms and neurotransmitter balance.

Anodal tDCS increases cortical excitability by depolarizing neurons, while cathodal tDCS decreases it through hyperpolarization. When combined with cognitive training, tDCS may produce faster and longer-lasting therapeutic effects. Although most of the neurorehabilitation studies have applied anodal excitatory stimulation, recent evidence suggests the potential cathodal inhibitory stimulation in neurodevelopmental disorders with alteration of synaptic transmission, as people with DS. Potentially both anodal and cathodal stimulation protocols could lead to positive clinical effects in DS.

This proof-of-concept study is a double-blind, placebo-controlled, clinical trial aiming to evaluate the efficacy of two active tDCS protocols (anodal and cathodal) targeting the left inferior frontal gyrus (IFG) versus sham stimulation tDCS, combined with speech and language training, to improve language skills in adolescents and young adults with DS. The study also aims to identify the most effective parameters of tDCS treatment, for customization in adolescents and young adults with DS. Thirty-six participants, aged 12 to 21 years, will be randomly assigned to three groups receiving anodal, cathodal, or sham tDCS. Each participant will undergo 10 sessions of tDCS at 1 mA for 20 minutes, alongside speech and language training five times for two weeks.

Neuropsychological, behavioral, biomarker (including brain-derived neurotrophic factor and neurofilament light chain), and electroencephalogram assessments will be performed at baseline, post-treatment, and three months after treatment completion. The study hypothesizes that tDCS will enhance language abilities, particularly expressive vocabulary, and modulate biomarkers of brain plasticity in DS participants. The study also hypothesizes that tDCS will enhance other cognitive and behavioral functions. Since tDCS effects may last, the study will check for improvements at the three-month. If effective, this combined approach of tDCS and language training could pave the way for new rehabilitation strategies for DS.

DETAILED DESCRIPTION:
Down Syndrome (DS), caused by trisomy 21, is the leading genetic cause of Intellectual Disability. This chronic and complex condition disrupts normal brain development and function, resulting in deficits in cognition and adaptive behavior. A hallmark of DS is cognitive impairment, characterized by low IQ and difficulties in learning, language processing, and executive functioning-largely associated with atypical neural organization.

In recent years, substantial progress has been made in uncovering the pathogenetic mechanisms responsible for these deficits. Research has identified specific neuroanatomical and neurochemical abnormalities, including alterations in the glutamatergic and GABAergic systems, as well as dysregulation of neuromodulators such as noradrenaline, dopamine, and acetylcholine. Individuals with DS also exhibit compromised synaptic plasticity, reduced neurogenesis, and diminished neural remodeling capacity-all contributing to their unique cognitive profile.

These neurobiological insights have spurred interest in developing therapeutic interventions aimed at improving cognitive function. Although some pharmacological strategies have shown promise in preclinical and limited clinical trials, their clinical translation has often yielded limited success, underscoring the need for alternative approaches. Among these, non-invasive brain stimulation (NiBS), particularly Transcranial Direct Current Stimulation (tDCS), is emerging as a promising method to enhance cognitive and language abilities.

The primary goal of this project is to build a robust scientific basis for novel brain-targeted rehabilitation strategies, specifically to address language deficits in adolescents and young adults with DS. Given the limited research on NiBS in this population, this proof-of-concept study aims to evaluate the feasibility and efficacy of two active tDCS protocols-anodal and cathodal stimulation-targeting the left inferior frontal gyrus (IFG), both compared to a placebo (sham) stimulation condition.

This is a proof-of-concept, non-profit, single-center, prospective, randomized, double-blind, placebo-controlled trial. Both participants and outcome assessors will be blinded to treatment allocation. Thirty-six participants with DS, aged 12 to 21 years, will be randomly assigned to three groups receiving anodal, cathodal, or sham (placebo) tDCS combined with speech and language training. The intervention comprises ten sessions of either anodal tDCS, cathodal tDCS, or sham (placebo) stimulation, delivered over two consecutive weeks (five sessions per week), in conjunction with a tailored speech and language training protocol. The stimulation intensity will be set at 1 mA for 20 minutes per session, each speech and language treatment session, administered by a trained speech therapist, will last 20 minutes structured in 10 minutes of motor planning/programming and 10 minutes addressing lexical, morphosyntactic, and functional language domains.

A neuropsychological, linguistic, behavioural and functional communication assessment will be will be carried prior to (baseline - T0), following the end of the treatments after two weeks (T1) and at 3 months after the end of treatment (T2), to evaluate potential long-lasting benefits. In addition to behavioral and cognitive measures, the study will explore biological markers of treatment response, specifically plasma levels of Brain-Derived Neurotrophic Factor (BDNF) and Neurofilament Light Chain (NfL), as well as EEG recordings, to evaluate neuronal plasticity changes after treatment. The primary outcome measure will be expressive vocabulary assessed by the Naming subtests of the Battery for the Assessment of Language in Children aged 4 to 12 years (BVL_4-12).

Secondary outcome measures will include:

Language and verbal skills:

* Articulation, Naming, Semantic Fluency, and Phonological Fluency subtests of the Battery for the Assessment of Language in Children aged 4 to 12 years (BVL_4-12)
* Inconsistency Task - 28 Italian words, based on the Inconsistency subtest of the DEAP (Diagnostic Evaluation of Articulation and Phonology).
* Intelligibility in Context Scale (ICS): Italian version, a parent-report scale widely validated worldwide, allowing caregivers to rate their child's functional speech intelligibility with different communicative partners.

Adaptive behavior and cognitive function:

-Adaptive Behavior Assessment System - Second Edition (ABAS-II), a questionnaire summarizing information on adaptive behavior and skills.

Verbal Span Task (VST), assessing verbal short-term memory by having the examiner read aloud five sequences of high-frequency disyllabic words at one word per second.

Behavioral assessment:

* Conners' Parent Rating Scales Long Version, Revised, (CPRS-R:L) widely used for screening ADHD and related symptoms.
* Child Behavior Checklist 6-18 (CBCL/6-18), a 113-item parent-report instrument designed to assess behavior and emotional problems in children.
* Aberrant Behavior Checklist (ABC), used to evaluate challenging behaviors.

Sleep disturbances:

-Sleep Disturbance Scale for Children (SDSC), a parent-report questionnaire to collect information on sleep disturbances in children and adolescents.

Quality of life and parental stress:

* Pediatric Quality of Life Inventory (PedsQL) , a brief measure of health-related quality of life.
* Parenting Stress Index 4 (PSI-4), exploring parental stress levels in the parent-child relationship.

Adherence to safety protocols will be ensured throughout the study, with side effects systematically monitored using a standardized questionnaire after each session and during the follow-up period.

Ultimately, this study seeks to generate high-quality evidence on the effectiveness of tDCS-compared to placebo-in enhancing language and cognitive outcomes in DS, while contributing to the identification of biomarkers predictive of individual responsiveness to neuromodulation-based interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Italian speakers participants of both genders with the presence of a free trisomy 21 documented by karyotyping
2. Adolescents and young adults from 12 to 21 years old
3. Mental age ≥ 4 years (as assessed by Leiter-3 at baseline)
4. Scores < 2 SD at the denomination subtest of BVL_4-12
5. Be comprehensible to closest relatives, at least in part, exhibiting consistent speech sounds mesured by Intelligibility in Context Scale (ICS): Italian (McLeod, Harrison, & McCormack, 2012) with a cut-off of 3.5
6. Informed consent/absent from each patient and Informed consent from their caregivers.

Exclusion Criteria:

1. The presence of any neurosensory deficits, such as hypoacusis or serious visual impairments
2. The presence of epilepsy, familiarity with epilepsy and major psychopathological disorders
3. Scores < 10 points at the denomination subtest of BVL_4-12
4. Ability to verbally imitate less that 7 of 10 words during an imitation screening task
5. Undergoing concomitant speech therapy or psychopharmacological therapy for cognitive or behavioral improvement.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Expressive Vocabulary | Assessments will be conducted at three time points: baseline (T0, day 1), immediately post-treatment (T1, day 10), and at follow-up (T2, three months).
  The primary outcome measure will be expressive vocabulary assessed by the Naming subtests of the Battery for the Assessment of Language in Children aged 4 to 12 years (BVL_4-12).

SECONDARY OUTCOMES:
Articulation, Semantic Fluency and Phonological Fluency | Assessments will be conducted at three time points: baseline (T0, day 1), immediately post-treatment (T1, day 10), and at follow-up (T2, three months)
  These subtests from the Battery for the Assessment of Language in Children aged 4 to 12 years (BVL_4-12) assess various language abilities: articulation evaluates the clarity of speech sounds; naming measures the ability to retrieve and produce the correct names of pictured objects; semantic fluency tests the capacity to generate words within a given category; and phonological fluency assesses the ability to produce words beginning with specific letters. Together, these measures provide a comprehensive evaluation of expressive language skills in participants.
Adaptive level | T0 (baseline, Day 1), T1 (post-treatment, Day 10), T2 (3-month follow-up, Day 90)
  Adaptive Behavior Assessment System - Second Edition (ABAS-II) Scale to obtain the parent's observations about the youth's behaviour and gives a complete overview of child and adolescent adaptive behaviours.
Psychopathological measure - behavioral and psychopathological aspects | T0 (baseline, Day 1), T1 (post-treatment, Day 10), T2 (3-month follow-up, Day 90)
  Conners' Parent Rating Scale - Revised, Long Form (CPRS-R:L). Questionnaire used parent's observations about the youth's behaviour and gives a complete overview of child and adolescent psychopathological disorders.The T scores of each scale of the questionnaire will also be evaluated.
Psychopathological measure - behavioural and emotional problems | T0 (baseline, Day 1), T1 (post-treatment, Day 10), T2 (3-month follow-up, Day 90)
  Child Behavior Checklist for Ages 6-18 (CBCL/6-18) Questionnaire assesses behavioural and emotional problems in children and young people aged 6-18 years.The T scores of each scale of the questionnaire will also be evaluated.
Health-related quality of life measure | T0 (baseline, Day 1), T1 (post-treatment, Day 10), T2 (3-month follow-up, Day 90)
  Pediatric Quality of Life Inventory (PedsQL) measuring health-related quality of life in healthy children and adolescents and those with acute and chronic health conditions. the raw scores of each scale (Physical , Emotional , Social , School) and the respective mean scores (Physical SC, Emotional Functioning ,Social Functioning , School Functioning), the physical index (T_Physical) , the psychosocial index (T_Psychosocial) and the mean total score (Total Score) of the questionnaire, will be evaluated.
Quality of sleep | T0 (baseline, Day 1), T1 (post-treatment, Day 10), T2 (3-month follow-up, Day 90)
  Sleep Disturbance Scale for Children (SDSC) Sleepiness inventory is used to obtain the parent's observations about sleep disorders in children in five subdomains.T scores of each scale will be evaluated.
Intelligibility | T0 (baseline, Day 1), T1 (post-treatment, Day 10), T2 (3-month follow-up, Day 90)
  Intelligibility in Context Scale (ICS). The ICS is a parent-report questionnaire, widely translated and extensively validated internationally, through which caregivers assess their child's functional speech intelligibility across seven different communication partners. This tool provides insight into how well the child's speech is understood in everyday social contexts
Parenting Stress Index | T0 (baseline, Day 1), T1 (post-treatment, Day 10), T2 (3-month follow-up, Day 90)
  Parenting Stress Index, Fourth Edition (PSI-4), is a validated instrument used to assess parental stress levels, specifically focusing on the parent-child relationship. It provides insight into the stresses experienced by parents in relation to their child.
Inconsistency | T0 (baseline, Day 1), T1 (post-treatment, Day 10), T2 (3-month follow-up, Day 90)
  Inconsistency Task - 28 Italian words, based on the Inconsistency subtest of the DEAP (Diagnostic Evaluation of Articulation and Phonology).
  This task evaluates speech inconsistency by assessing participants' ability to produce consistent pronunciations of a set of 28 high-frequency Italian words.
Verbal Span | T0 (baseline, Day 1), T1 (post-treatment, Day 10), T2 (3-month follow-up, Day 90)
  Verbal Span Task (VST) assesses short-term verbal memory. During the task, the examiner reads aloud five sequences of high-frequency disyllabic words at a rate of one word per second, and participants are required to recall them.
Assessment of Challenging Behaviors | T0 (baseline, Day 1), T1 (post-treatment, Day 10), T2 (3-month follow-up, Day 90)
  The Aberrant Behavior Checklist (ABC) is a standardized questionnaire designed to assess challenging behaviors in individuals with developmental disabilities. It evaluates domains such as irritability, aggression, hyperactivity, lethargy, and social withdrawal, providing a comprehensive profile of maladaptive behaviors for clinical and research purposes.

OTHER OUTCOMES:
Biological measures | T0 (baseline, Day 1), T1 (post-treatment, Day 10), T2 (3-month follow-up, Day 90)
  The evaluation of Brain-Derived Neurotrophic Factor (BDNF) and Neurofilament Light Chain (NfL) levels is performed through the collection of blood samples.
  Blood samples will be collected by venipuncture between 8 and 10 pm at baseline (T0), at the end of treatment (T1) and after three months (T2). Plasma levels of BDNF and NfL will be measured by enzyme-linked immunosorbent assay (ELISA) according to the procedures supplied by the manufacturer (DuoSet, R&D Systems, Minneapolis, MN, USA). Analyses of blood samples were also performed blind to group assignment and outcome. The BDNF content and the NfL will be measured on plasma samples obtained from 7 cc blood collected in EDTA tubes, centrifuged at 1000 x g for 15 min, and immediately stored at -20°C avoiding repeated freeze-thaw cycles.
Neurophysiological measures | T0 (baseline, Day 1), T1 (post-treatment, Day 10), T2 (3-month follow-up, Day 90)
  Electroencephalogram (EEG) is a method to record an electrogram of the electrical activity on the scalp that has been shown to represent the macroscopic activity of the surface layer of the brain underneath. Resting-state EEG will be recorded in a sound-attenuated, electrically shielded room through a 8-channels positioned close to the region of interest (IFG), reusable pre-wired headcap system to minimize preparation time. Participants will be instructed to sit comfortably and relax. A minimum time of 5-minutes EEG activity with eyes closed will be recorded. EEG signals will be amplified at a sampling rate of 1000 Hz using a 0.1-100 Hz online bandpass filter. For each channel, a 0.5-45 Hz offline, digital bandpass filter will be applied, and electrode impedance will be kept below 50 k omega. To reduce artifacts, Curry 7 will be used for EEG data pre-processing.

CONTACTS AND LOCATIONS:
Locations (1):
- Bambino Gesù Children's Hospital, IRCCS, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopes JBP, Grecco LAC, Moura RCF, Lazzari RD, Duarte NAC, Miziara I, Melo GEL, Dumont AJL, Galli M, Santos Oliveira C. Protocol study for a randomised, controlled, double-blind, clinical trial involving virtual reality and anodal transcranial direct current stimulation for the improvement of upper limb motor function in children with Down syndrome. BMJ Open. 2017 Aug 11;7(8):e016260. doi: 10.1136/bmjopen-2017-016260. PMID 28801420
- [Background] Lopes JBP, Miziara IM, Kahani D, Parreira RB, de Almeida Carvalho Duarte N, Lazzari RD, Santos LV, de Mello Monteiro CB, da Silva Cardoso DC, de Oliveira Hassel Mendes J, Dos Santos Alves VL, Silva IO, Oliveira LV, Conway BA, Galli M, Cimolin V, Oliveira CS. Brain activity and upper limb movement analysis in children with Down syndrome undergoing transcranial direct current stimulation combined with virtual reality training: study protocol for a randomized controlled trial. Trials. 2022 Jan 28;23(1):87. doi: 10.1186/s13063-022-06014-4. PMID 35090554
- [Background] Faralli A, Fuca E, Lazzaro G, Menghini D, Vicari S, Costanzo F. Transcranial Direct Current Stimulation in neurogenetic syndromes: new treatment perspectives for Down syndrome? Front Cell Neurosci. 2024 Feb 22;18:1328963. doi: 10.3389/fncel.2024.1328963. eCollection 2024. PMID 38456063
- See also: Study information brochure approved. — https://specchioriflesso.net/media/213835/brochure_informativa_cartacea_versione_1.0_17_06_2024.pdf